CLINICAL TRIAL: NCT06885606
Title: Using Transcranial Direct Current Stimulation (tDCS) for Vaping Reduction in Daily E-cigarette Users: a Pilot Study
Brief Title: The Use of TDCS for Vaping Reduction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Senior Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 007/2023
Record Dates: First submitted 2023-12-19; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Vaping; Addiction; Transcranial Direct Current Stimulation(tDCS)
Keywords: E-cigarettes; Vaping; Brain stimulation; tDCS; Nicotine
MeSH Terms: conditions — Vaping; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active tDCS stimulation group (Active Comparator)
  Interventions: Device: Active tDCS
- Sham tDCS stimulation group (Sham Comparator): Sham tDCS applies a 2mA current for the initial 30 seconds, followed by 0 mA for the remaining 19.5 minutes to simulate active tDCS stimulation. The cathode electrode is placed on the right dorsolateral prefrontal cortex (DLPFC), and the anode is positioned on the left DLPFC, aligned with the electrode placement used in active tDCS.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Active tDCS — Transcranial direct current stimulation (tDCS) is a form of non-invasive brain stimulation that involves brief (e.g., 20-min) application of weak electric current (e.g., 2 mA) to the scalp. Active tDCS intervention increases excitability of neurons at the anode with 20-30% of the current going through the brain from anode to cathode so that both cortical and subcortical structures are stimulated. The procedure is very safe, convenient, and fast-acting with well-established parameters. It has the ability to modulate plasticity in specific brain areas and has established efficacy in human laboratory models of addictive motivation and has been shown to decrease craving for cigarettes when the anode is placed over the left dorsolateral prefrontal cortex (DLPFC).
  Arms: Active tDCS stimulation group
Device: Sham tDCS — Sham tDCS applies a 2mA current for the initial 30 seconds, followed by 0 mA for the remaining 19.5 minutes to simulate active tDCS stimulation. The cathode electrode is placed on the right dorsolateral prefrontal cortex (DLPFC), and the anode is positioned on the left DLPFC, aligned with the electrode placement used in active tDCS.
  Arms: Sham tDCS stimulation group

SUMMARY:
Project Summary - tDCS for Vaping Reduction

Background: While the prevalence of tobacco smoking has plateaued over the last several years, the prevalence of nicotine vaping (e-cigarettes) continues to increase exponentially in Canada. Originally touted as a safe alternative to smoking, e-cigarette use or vaping is now most popular among youth and young adults. The high prevalence of e-cigarette use, coupled with growing evidence of associated harms and reports of addiction and difficulties in quitting reinforces the urgent need to develop and test methods to attenuate e-cigarette craving as a step towards developing approaches to vaping cessation that are brief, inexpensive and effective. Non-invasive brain stimulation techniques have become a popular area of research as a treatment option for substance use disorders with growing evidence of their effectiveness for a variety of addictions. One of these techniques, transcranial direct current stimulation (tDCS), has been shown to decrease cigarette craving and consumption. Thus, the purpose of this pilot study is to evaluate the effectiveness of using tDCS for vaping reduction in e-cigarette users.

Methods: This will be a double-blind sham-controlled randomized trial whereby 40 daily nicotine-containing e-cigarette users will be recruited to undergo 10 consecutive daily sessions of tDCS (Monday to Friday for 2 weeks). Participants will be randomized (1:1) to either sham (0mA) or active tDCS (2mA), with the anode at the left dorsolateral prefrontal cortex (DLPFC) and cathode at the right DLPFC. The primary outcome is vaping frequency (puffs/day and nicotine pods/week) at end of treatment (2 weeks). The secondary outcome will be e-cigarette craving. Participants will be followed-up via the phone at 1 month and 3 months post randomization respectively.

Implication: This will be the first treatment study to target vaping reduction. There are currently no established treatment options for e-cigarette addiction and medications traditionally used for smoking cessation only address withdrawal symptoms and not addiction pathology. Thus, findings from this study may be used to inform future designs of vaping reduction strategies or vaping cessation.

ELIGIBILITY:
Inclusion Criteria:

* The participant must meet all of the inclusion criteria to be eligible for this research study:

  1. Be able to provide informed written consent
  2. Stated willingness to comply with all study procedures
  3. Age 18 - 65 years
  4. Is a daily regular use of nicotine-containing e-cigarette for at least the past 6 months
  5. Is willing to attend daily appointments for tDCS for two consecutive weeks (Monday through Friday)
  6. Is not interested in or planning to quit vaping in the next 30 days.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this research study:

  1. Substance use disorder (other than nicotine dependence) (M.I.N.I. SCID) (confirmed with urine drug screen)
  2. Current regular use of tobacco cigarettes, nicotine replacement therapy or other medications for smoking cessation
  3. Unstable psychiatric condition
  4. Recent clinically significant head trauma*
  5. History of seizures and/or epilepsy*
  6. Pacemakers or implanted electrical devices such as cochlear implants*
  7. Metal embedded in the skull*
  8. Skin lesions, open wounds, bruising, or similar injuries on the scalp*

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Explore the efficacy of tDCS for reducing vaping use. | 2 weeks
  The primary outcome is frequency of vape use at end of treatment (2 week period), measured by self-reported vaping frequency (puffs/day) and nicotine pods/week (estimate total nicotine consumed per week).

SECONDARY OUTCOMES:
Explore changes in craving that are associated with tDCS intervention. | 2 weeks
  The secondary outcome of this study will be e-cigarette craving at end of treatment (2 week period), as well as vaping use at 3 months follow up.

IPD SHARING:
Plan to Share IPD: No